CLINICAL TRIAL: NCT02003443
Title: Acupressure for the Treatment of Pain in Older Adults With Symptomatic Knee Osteoarthritis
Brief Title: Acupressure for Knee Pain in Older Adults
Acronym: AKP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lydia W Li, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N015749; 5968 (Other Grant/Funding Number: Arthritis Foundation)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis
Keywords: Acupressure; Older Adults; Knee pain; Pain Treatment
MeSH Terms: conditions — Osteoarthritis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham Acupressure (Placebo Comparator): Participants assigned to sham acupressure will receive similar instruction as those assigned to pain-relief acupressure, except that they will be taught to apply pressure to 10 acupoints that are unrelated to pain. That is, they will conduct self-administered acupressure 5 days/week for 8 weeks, as the pain-relief acupressure group does, but on 'sham' acupoints.
  Interventions: Behavioral: Self-Administered Acupressure
- Usual Care (No Intervention): Participants assigned to the UC group will receive no intervention.
- Pain-Relief Acupressure (Experimental): Participants assigned to pain-relief acupressure will be taught to apply physical pressure, using a wooden hand-held device designed for acupressure, to 10 acupoints on their body.That is, they will conduct self-administered acupressure 5 days/week for 8 weeks,on acupoints that are relevant to pain reduction.
  Interventions: Behavioral: Self-Administered Acupressure

INTERVENTIONS:
Behavioral: Self-Administered Acupressure — The intervention involves teaching and supporting subjects to administer acupressure on themselves.
  Arms: Pain-Relief Acupressure; Sham Acupressure

SUMMARY:
The primary objective of this project is to determine whether self-administered acupressure is an effective and feasible self-management strategy for older adults with symptomatic KOA. Participants will be randomized to three treatment groups: pain-relief acupressure, sham acupressure, and usual care (UC). The two acupressure groups will be taught to administer pain-relief and sham acupressure, respectively, on themselves 5 days/week for 8 weeks. The usual care group will not be required to change any of their treatment practice. Outcome data will be collected at baseline, and the 4th and 8th week after baseline.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a leading cause of disability in the elderly and this disability is commonly attributed to knee pain. Current treatments for knee pain are only modestly efficacious, and some common treatments like non-steroidal anti-inflammatory drugs (NSAIDS) have adverse long-term effects. Acupressure is an inexpensive and noninvasive treatment that has the potential to be a useful long-term self-management strategy for pain. Acupressure can be easily taught and is safe enough to self-apply without supervision. Participants will be randomized to three treatment groups: pain-relief acupressure, sham acupressure, and usual care (UC). The intervention will last for 8 weeks during which participants in the pain-relief and sham acupressure groups will be taught the assigned treatment by a trained research assistant who is blinded to the treatment arm, and provided with a digital video disc to aid their practice at home. The UC group will not receive training from the research team or be required to change their treatment practice.Our research team will make weekly phone calls to all three groups of participants to ask about their pain levels and any adverse events. For the two acupressure groups, the phone calls serve to support the participants' adherence to treatment. Data will be collected at baseline, mid-point (4 weeks after baseline) and the end ( 8 weeks) of the intervention. These results will help us assess the efficacy of pain-relief acupressure on knee pain in older adults, and allow us to calculate effect sizes to determine the appropriate sample size for a larger future study. Since no studies have involved older adults in self-administered acupressure, information about feasibility of and adherence to using this method in older adults would be invaluable.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Community-living (i.e., own home, senior residence, apartment)
* Have a physician diagnosis of knee OA
* Current persistent pain (pain ≥ 4 on a 1-10 Visual Analogue Scale on 50% or more of days) that has lasted for 3 months or longer
* Ability to speak and write in English
* Adequate cognitive status (score > 5 on the 6-item screener)
* Adequate functional ability to administer the acupressure protocol (e.g., able to use fingers or device to apply pressure to acupoints, able to easily reach feet to access acupoints)
* Ability to demonstrate understanding of treatment protocol through demonstration after being instructed
* Ambulatory with or without an assistive device
* Adequate hearing and vision to follow study protocol
* Agree not to start any new therapy for pain control during the study period
* Have a telephone and television

Exclusion Criteria:

* Receiving active cancer treatment
* Have a bleeding diathesis condition
* Have health conditions that could confound the effect of acupressure (e.g., rheumatoid arthritis, lupus, diabetic neuropathy)
* Had knee replacement surgery
* Planned or current involvement in physical therapy, acupuncture or acupressure during the study period or receipt of any of these in the previous 3 months
* Knee injection in prior 6 weeks with no planned injection during the study period
* Chronic use of opioid therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pain | 4 and 8 Weeks
  The Western Ontario McMaster Universities Osteoarthritis Index (WOMAC).

SECONDARY OUTCOMES:
Physical Function | 4 and 8 weeks
  Both objective and subjective assessments of physical function will be used. The 6 minute walk and the timed up and go (TUG) tests are the objective measures. The 6 minute walk test has been demonstrated to yield reliable measurements of exercise capacity and is frequently used in OA trials. The TUG is a test of functional ability and measures the time (in seconds) to get up from a chair, walk 20 feet and return to the chair. For subjective assessment, we will use the physical function subscale (17 items) of WOMAC.

OTHER OUTCOMES:
Fatigue | 4 and 8 weeks
  Fatigue will be measured by the Brief Fatigue Inventory (BFI).

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Li, PhD, Principal Investigator — Regents of the University of Michigan
Locations (1):
- University of Michigan Chronic Pain and Fatigue Research Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Li LW, Harris RE, Tsodikov A, Struble L, Murphy SL. Self-Acupressure for Older Adults With Symptomatic Knee Osteoarthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Feb;70(2):221-229. doi: 10.1002/acr.23262. Epub 2017 Dec 29. PMID 28437570